CLINICAL TRIAL: NCT01001858
Title: Domiciliary Diagnosis and Follow up in Obstructive Apnoea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Ada Luz Andreu Rodríguez, HOspital San Juan de Alicante. España
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7387
Record Dates: First submitted 2009-10-07; First posted 2009-10-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; CPAP compliance; nurse domiciliary led; sleep disease
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Domiciliary group (Active Comparator): In this group OSA diagnosis was performed at patient's home by mean of non-attended RP. All follow-up visits were conducted by a trained nurse in patient's home.
  Interventions: Other: Diagnosis and monitoring of OSA patients
- Hospital Group (Active Comparator): In this group diagnosis was made by in-hospital PSG. Follow-up was performed at hospital by a specialist Physician
  Interventions: Other: Diagnosis and monitoring of OSA patients
- Mixed Group (Active Comparator): In this group diagnosis was made by home RP, and follow-up at hospital
  Interventions: Other: Diagnosis and monitoring of OSA patients

INTERVENTIONS:
Other: Diagnosis and monitoring of OSA patients — The difference between the three strategies is given by the method used for OSA diagnosis (domiciliary RP or hospital PSG) and the type of monitoring carried out after initiating CPAP treatment (by physician at hospital or by a trained nurse in patient's home)
  Other Names: Domiciliary group: group A; Hospital group: group B; Mixed Group: groupC

SUMMARY:
The aim of the investigators study was to evaluate the effectiveness of a home programme (diagnosis and follow-up) in patients with Obstructive Sleep Apnea (OSA) syndrome treated with CPAP and to analyze the cost of this approach.

DETAILED DESCRIPTION:
The aim of our study was to evaluate the effectiveness of a home programme (diagnosis and follow-up) in patients with Obstructive Sleep Apnea (OSA) syndrome treated with CPAP and to analyze the cost of this approach.

Detailed Description: We conducted a prospective comparative study. Patients referred for suspected OSAS were evaluated. In the first visit patients completed four questionnaires: Epworth sleepiness scale, Impact Functional Illness Questionnaire (FOSQ), activity questionnaire and symptom questionnaire.

Patients were randomised to three groups:

* Group A (domiciliary group): home based diagnosis by home respiratory polygraphy (RP) and home review conducted by a specialist nurse
* Group B (Hospital group): hospital based diagnosis by polysomnography (PSG) and clinical review conducted by a Pulmonologist
* Group C (mixed group): home based diagnosis by home respiratory polygraphy (RP) and clinical review conducted by a Pulmonologist

Following the diagnostic test (PSG or RP), patients were visited by the Pulmonologist, who identified the need for CPAP treatment.

Patients were evaluated after 1,3 and 6 months of CPAP treatment. In all follow-up visits compliance was evaluated by objective methods and questionnaires described above were filled in.

In domiciliary group, phone calls or hospital appointments were made if low compliance was detected or if some problem with treatment was detected.

Instrumentation.

* Conventional PSG was performed in hospital supervised by a trained nurse. PSG used for the study was Somnostar alfa®. Parameters obtained were: electroencephalogram (C3-A2, C4-A1), electrooculogram electromyogram, electrocardiogram (V2 modified), respiratory effort by thoracic and abdominal resistance bands, air flow with nasal cannula pressure connected to a transducer, oxygen saturation with a pulseoximeter, and snoring with a selective microphone. PSG was manually interpreted in 30 seconds epochs, according to Rechschaffen and Kales criteria.The apnea-hypopnea index (AHI) was defined as the number of apneas-hypopneas divided by the number of hours of sleep. OSA diagnosis was done if AHI was >10 /h.
* Respiratory polygraphy was performed in a non-attended way in patient's home. The nurse who monitorized the patient in the home setting, instructed the patient on the proper use of the RP. A validated respiratory polygraphy system corresponding to ASDA level III (Stardust®) was used. The parameters monitorized were: nasal flow, chest movement, oxyhemoglobin saturation, pulse and body position. The same cardio-respiratory variables that we identified in PSG, were registered. An event rate (number of apneas + number of hypopnea divided by the number of hours recorded)> 15 was considered as a diagnosis. The study were recorded by computer system and manually interpreted by a physician. In case of invalid registration we performed a second PR. If in doubt after the second study a PSG was performed.

Follow-up visits and assessment of compliance:

* Hospital monitoring group: Effective compliance was calculated by mean of the CPAP hour meter, dividing the total number of hours timer by the number of days of use. We discounted 10% of the time, which is the average time of ineffective pressure. Patients were considered adherent if they use CPAP at least 4 hours during 70% of the week
* Follow-up visits by nurses: This group of patients was treated at home through a system of fixed pressure CPAP (REMstar Pro, Respironics ®), with a memory card which can store information about the number of hours of effective pressure. It also allows to know the number of days of CPAP use. In all visits the nurse collect the memory card for later analysis, which was performed by a physician.The nurse responsible for the program evaluated the need of reinforcing in order to get an optimal compliance. If it was considered necessary, the patient was evaluated by the Pulmonologist either by mean of a phone call or of an hospital appointment. All patients in this group were contacted by phone at least once during the first month of CPAP treatment

ELIGIBILITY:
Inclusion criteria:

Patients with high probability of OSA, defined by two or more of :

* daytime sleepiness
* snoring
* recognized apnoeic episodes
* associating obesity and / or hypertension

Exclusion Criteria:

* Patients with impaired lung function ( overlap syndrome, obesity-hypoventilation syndrome, restrictive disorders), associated pathology (psychiatric disorder, periodic limb movements, dyssomnias or other parasomnias)
* Patients treated with CPAP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Differences in compliance among the three different strategies, measured by CPAP hours of use | six months follow-up

SECONDARY OUTCOMES:
costs of the three different strategies, including number of visits and phone calls that were necessary to improve compliance and additional diagnostic tests. | six months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eusebi Chiner Vives, MD, Study Director — Jefe de Sección de Neumología del Hospital San Juan de Alicante. España
Locations (1):
- Hospital San Juan de Alicante, San Juan, Alicante, Spain

REFERENCES:
- [Derived] Andreu AL, Chiner E, Sancho-Chust JN, Pastor E, Llombart M, Gomez-Merino E, Senent C, Barbe F. Effect of an ambulatory diagnostic and treatment programme in patients with sleep apnoea. Eur Respir J. 2012 Feb;39(2):305-12. doi: 10.1183/09031936.00013311. Epub 2011 Jun 30. PMID 21719490